CLINICAL TRIAL: NCT02220816
Title: Efficacy of an Attentional Process Training Using Competitive Versus Non Competitive Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Nisa (Other)
Collaborators: Universitat Politècnica de València (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NISA-COG-2014/1
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Stroke; Brain Injuries
Keywords: Attention; Competitive; Training
MeSH Terms: conditions — Stroke; Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Competitive Training (Experimental): The patients will receive only competitive activities designed to restore attention abilities. These include pencil-and-paper tasks completed under competitive circumstances and competitive virtual games specifically designed to treat different aspects of attention (divided, selective, sustained, etc).
  Interventions: Behavioral: Competitive training
- Non-Competitive Training (Active Comparator): The patients will receive conventional attentional training. Pencil and paper tasks focused on different aspects of attention (divided, selective, sustained, etc.) will be completed by all participant under individual or group-therapy sessions. No competitive training will be allowed.
  Interventions: Behavioral: Non-Competitive Training

INTERVENTIONS:
Behavioral: Competitive training — 30 sessions of competitive cognitive training; 3 - 5 sessions/week; duration 45 min
  Arms: Competitive Training
Behavioral: Non-Competitive Training — 30 sessions of non-competitive cognitive training; 3 - 5 sessions/week; duration 45 min
  Arms: Non-Competitive Training

SUMMARY:
Within a prospective, randomised, controlled study 60, selected patients with chronic (> 6 months) stroke or traumatic brain injury will be randomised to 30 1-hour sessions of competitive versus non-competitive attentional training. Competitive training will include fifteen 1-hour sessions of standard (paper and pencil) training under competitive situations and fifteen 1-hour sessions of competitive attentional games designed for this purpose using a new virtual reality system (conventional liquid-crystal-display screen with an infrared LED array to facilitate multi-touch experience embedded in a conventional table). Progress will be evaluated by pre and post measurement of attentional neuropsychological tests, subjective reports of global attention, usability and motivational scales. Our hypothesis is that competitive training is more effective in improving attention than conventional training in the chronic phase after acquired brain injury.

DETAILED DESCRIPTION:
Participants: Sixty 18-75 years-old patients with acquired brain injury, will be randomly assigned to 30 sessions of competitive versus non-competitive cognitive attentional training (see inclusion-exclusion criteria). Material and Methods: Randomized clinical trial comparing two different attentional training strategies. Attentional measures, usability data and caregiver/family perception of change, will be compared after completing both conditions. Competitive training will include a new computer based training program that involve using attentional skills under different competitive scenarios. Attentional exercises were designed according to the instructions of two experts neuropsychologists and included game-based situations simulating different olympic disciplines.Neuropsychological protocol: An assessment before the beginning of the intervention and pos-treatment will be done by a trained blinded neuropsychologist using measures of selective, sustained, divided and alternating attention (see primary outcome measures). Usability and Motivation: It is well-known that game-based cognitive exercises can increase motivation to treatment which in turn can increase learning strategies and improve outcomes after rehabilitation processes. Competitive tasks can also improve the effort and interest of the players and the intensity of the task through increasing motivation to win, get a reward and beat the others. Since motivation was an important element of our research, we assessed this capacity at the end of the treatment with the Intrinsic Motivation Scale. Also, the revised Competitiveness Index was used to measure the subject's preference for competitive situations. Finally, usability was considered a secondary outcome of our study since most of the games employed here were designed to be played in a new virtual reality system which was build to facilitate competitive strategies among 2-4 players (see secondary outcomes). Sample Size Calculation: There was any previous study that used the design proposed in this investigation. Considering a reduction bigger of 20% on the Hit-Reaction Time of the CPT-II scores in the active group intervention, sample size in both groups of 27 participants and standard-deviation in the magnitude of half of the medium score in each group (moderate variability), the study will be able to detect a moderate effect size (ES = 0,4). Calculating a sample loss of 10% each group, we define a sample size per group of 30 individuals. Statistical methods Statistical analyses will be performed with Statistical Package for the Social Sciences (SPSS) 12.0. The univariate analyses will be performed with the t student test / Mann-Whitney to continuous variables or Chi-Square test (X²) / Fischer test to categorical variables. The effective of the intervention over time will be assess through analyses of mixed models (repeated measures ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Acquired brain injury patients (stroke and traumatic brain injury)
* Chronicity > 6 months
* More than 3 months under cognitive rehabilitation
* Mississippi Aphasia Screening Test (comprehension subtest > 45)

Exclusion Criteria:

* Severe cognitive impairment defined as < 23 on Mini Mental Status Examination
* Unable to give informed consent
* Visual or auditive disorders limiting the ability to comply with treatment regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in attentional psychometric measures | Baseline versus end of treatment (an expected average of 8 weeks)
  Neuropsychological battery: Conner's Continuous Performance Test (CPT-II), Color-Trail Test, d2, Stroop test, Wechsler Adult Intelligence Scale-IV digit-span, Corsi block-tapping test

SECONDARY OUTCOMES:
Usability measures | Baseline versus end of treatment (an expected average of 8 weeks)
  System Usability Scale, Intrinsic Motivation Inventory

OTHER OUTCOMES:
Family-centered outcomes | Baseline versus end of treatment (an expected average of 8 weeks)
  Moos Attention Rating Scale, Subjective perception of improvement

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Llorens, PhD, Principal Investigator — Universitat Politècnica de València
Locations (1):
- Hospitales NISA, Valencia, Valencia, Spain